CLINICAL TRIAL: NCT05130437
Title: A Phase 1/2, Global, Open-Label, Extension Study to Evaluate the Long-Term Safety and Clinical Activity of mRNA-3927 in Participants Previously Enrolled in the mRNA-3927-P101 Study
Brief Title: A Study to Assess the Long-term Safety and Clinical Activity of mRNA-3927 in Participants Previously Enrolled in the mRNA-3927-P101 Study
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: mRNA-3927-P101-EXT; 2022-502911-12-00 (Other: Clinical Trials Information System (CTIS))
Record Dates: First submitted 2021-11-03; First posted 2021-11-23 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Propionic Acidemia
Keywords: mRNA-3927; Propionic Aciduria; Metabolism, Inborn Errors; Genetic Diseases; Inborn Amino Acid Metabolism, Inborn Errors; Acidosis; Acid-Base Imbalance; Metabolic Diseases; Organic Acidemias; Moderna; mRNA
MeSH Terms: conditions — Propionic Acidemia; Metabolism, Inborn Errors; Genetic Diseases, Inborn; Amino Acid Metabolism, Inborn Errors; Acidosis; Acid-Base Imbalance; Metabolic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- mRNA-3927 (Experimental): Participants will receive the applicable dose identified during Study mRNA-3927-P101 (NCT04159103) on Day 1. The dose can be adjusted based on Sponsor recommendation.
  Interventions: Biological: mRNA-3927

INTERVENTIONS:
Biological: mRNA-3927 — mRNA-3927 dispersion for IV infusion

SUMMARY:
The main purpose of this study is to evaluate the long-term safety of mRNA-3927 administered to participants with propionic acidemia (PA) who have previously participated in Study mRNA-3927-P101 (NCT04159103).

DETAILED DESCRIPTION:
The study will assess long-term safety of mRNA-3927. Participants with PA who were previously enrolled and completed the end-of-treatment (EOT)/early termination (ET) visit of the mRNA-3927-P101 study will have the option to enroll into this extension study provided all eligibility criteria have been met.

The study will include 2 periods: 1) Treatment Period and 2) Follow-up Period (90 days after the EOT visit). All participants will enter the study receiving mRNA-3927 at the same dose and at the same dosing interval last received in the mRNA-3927-P101 study.

ELIGIBILITY:
Inclusion Criteria:

* Participated in Study mRNA-3927-P101.
* Completed the EOT/ET visit in Study mRNA-3927-P101 and enroll in this study such that the first dose in this study is planned to be within 14±3 days of the last dose of mRNA-3927 in the mRNA-3927-P101 study.

Exclusion Criteria:

* Not expected to receive clinical benefit from continued mRNA-3927 administration, in the opinion of the Investigator.
* Any clinical or laboratory abnormality or medical condition that, at the discretion of the Investigator, may put the individual at increased risk by participating in this study.
* History of liver and/or kidney transplant.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-11-09 (Actual); Primary Completion 2029-12-04 (Estimated); Study Completion 2031-12-04 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs), Serious AEs (SAEs), and AEs Leading to Discontinuation | Baseline through End of Study Visit (up to 8 years)

SECONDARY OUTCOMES:
Annualized Frequency of Investigator-reported Metabolic Decompensation Events (MDEs) | Baseline through End of Study Visit (up to 8 years)
Annualized Frequency of Investigator-reported MDE-related Hospitalizations | Baseline through End of Study Visit (up to 8 years)
Annualized Frequency of Investigator-reported PA-related Hospitalizations | Baseline through End of Study Visit (up to 8 years)
Annualized Frequency of Investigator-reported PA-related Urgent Healthcare Encounters | Baseline through End of Study Visit (up to 8 years)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (6):
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - University of Michigan Hospitals, Ann Arbor, Michigan
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Duke University Medical System (Duke Health), Durham, North Carolina
  - The Children's Hospital of Philadelphia (CHOP), Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
- Hospital For Sick Children, Toronto, Ontario, Canada
- Fujita Health University Hospital, Toyoake-shi, Akita, Japan
- United Kingdom (4):
  - Willink Biochemical Genetics Unit - Manchester, Manchester, England
  - University Hospital Birmingham NHS Foundation Trust, Birmingham, West Midlands
  - Birmingham Women's and Children's NHS Foundation Trust, Birmingham, West Midlands
  - Great Ormond Street Hospital for Children NHS Foundation Trust, London